CLINICAL TRIAL: NCT07194200
Title: Evaluating the Safety and Efficacy of Lactobacillus Plantarum in Treating Psoriasis: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Safety and Efficacy of Lactobacillus Plantarum for Psoriasis: A Randomized Double-Blind Placebo-Controlled Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LL-KY-2025150-02
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis; Lactobacillus Plantarum
Keywords: psoriasis; Lactobacillus plantarum
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: Intervention measures for the experimental group: Apply 5ml of Lactobacillus plantarum solution extracted from the skin surface of healthy individuals to the psoriatic lesions daily, for a duration of 2 months.
  Intervention measures for the control group: Apply 5ml of inactivated Lactobacillus plantarum solution to the psoriatic lesions daily, for a duration of 2 months.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Experimental): Intervention measures for the experimental group: Apply 5ml of Lactobacillus plantarum solution extracted from the skin surface of healthy individuals to the psoriatic lesions daily, for a duration of 2 months.
  Interventions: Biological: Lactobacillus plantarum
- group B (Active Comparator): Intervention measures for the control group: Apply 5ml of inactivated Lactobacillus plantarum solution to the psoriatic lesions daily, for a duration of 2 months.
  Interventions: Biological: inactivated Lactobacillus plantarum

INTERVENTIONS:
Biological: Lactobacillus plantarum — Intervention measures for the experimental group: Apply 5ml of Lactobacillus plantarum solution extracted from the skin surface of healthy individuals to the psoriatic lesions daily, for a duration of 2 months.
  Arms: group A
Biological: inactivated Lactobacillus plantarum — Intervention measures for the control group: Apply 5ml of inactivated Lactobacillus plantarum solution to the psoriatic lesions daily, for a duration of 2 months.
  Arms: group B

SUMMARY:
A growing body of evidence indicates that the pathogenesis of psoriasis may be closely linked to skin microbiome dysbiosis. Compared with healthy individuals, the composition and function of the skin microbiota in psoriasis patients exhibit significant alterations5,6. This microbial imbalance is thought to contribute to the initiation and progression of the disease through mechanisms such as triggering abnormal immune responses, exacerbating inflammatory processes, and impairing the skin barrier.

In-depth exploration of the interplay between psoriasis and the microbiome not only offers new perspectives for elucidating the disease's pathogenesis but also lays the groundwork for developing innovative microbiota-targeted diagnostic and therapeutic strategies. Thus, identifying novel therapeutic approaches that bridge psoriasis treatment and microbial regulation holds substantial clinical and social value.

While existing treatments for psoriasis have made some progress, research specifically focusing on the microbiota-psoriasis relationship remains relatively limited. Investigating the intrinsic connections between microecological balance and psoriasis management, and developing practical improvement strategies, is therefore of crucial practical significance for enhancing skin health and improving quality of life. This study aims to address this research gap and provide a new therapeutic option for individuals with psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Reference to Psoriasis Area and Severity Index (PASI) score < 10 Patients have been informed of the study details, voluntarily participate, and have signed the informed consent form; Aged 18-60 years with good general health status; No use of any medications within 6 months; No various inflammatory or immune skin diseases, no local infections, and no neuromuscular diseases.

Exclusion Criteria:

* Patients with other types of psoriasis or severe psoriasis; Those in the active phase of skin diseases or with other serious diseases; Other situations deemed unsuitable for enrollment by the researchers, such as subjects who are untrustworthy, unable to accept or understand the study assessments.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Transepidermal Water Loss(TEWL) | The follow-up periods are set at 1, 2, 4, and 8 weeks after the initial treatment.
  Use a dermatological detector to measure the TEWL of the skin. Gently press the probe against the subject's skin, and the TEWL at that location will be displayed on the device's screen.
General appearance photography | The follow-up periods are set at 1, 2, 4, and 8 weeks after the initial treatment.
  After shooting, three professional doctors will independently assess the improvement of psoriatic lesions in patients.
Dermoscopic photography | The follow-up periods are set at 1, 2, 4, and 8 weeks after the initial treatment.
  After shooting, three professional doctors will independently assess the improvement of psoriatic lesions in patients.
Completion of self-assessment questionnaires | The follow-up periods are set at 1, 2, 4, and 8 weeks after the initial treatment.
  Record the improvement of patients' self-perceived suboptimal skin conditions after treatment compared with the baseline.
Adverse reactions | The follow-up periods are set at 1, 2, 4, and 8 weeks after the initial treatment.
  Subjects will record predefined expected post-treatment events at the treated sites.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No